CLINICAL TRIAL: NCT06217341
Title: Bispectral Index and Emergence Agitation in Spinal Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ahmet YUKSEK, Associate professor, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2023-32
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia Recovery Periods; Anesthesia Complication; Electroencephalography
Keywords: anesthesia; bispectral index; emergence agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- emergence agitation group: Patients in the emergence agitation group are patients who are observed to be agitated during recovery according to the Richmond agitation sedation scale after anesthesia.
  Interventions: Other: In the study, bispectral index monitoring and follow-up will be applied to both groups.
- calm group: The calm group will consist of patients whose agitation scale is below +2 during recovery.
  Interventions: Other: In the study, bispectral index monitoring and follow-up will be applied to both groups.

INTERVENTIONS:
Other: In the study, bispectral index monitoring and follow-up will be applied to both groups. — Perioperative Bispectral Index Monitoring (BIS) monitor and Bispectral Index suppression Rate (BIS-SR) monitoring will be applied. The duration and magnitude of BIS-SR values will be examined together with BIS values in terms of recovery agitation.
  Other Names: Bispectral Index Monitoring

SUMMARY:
Recovery and emergence agitation is a problem that occurs after anesthesia and requires urgent intervention. The effects of changes in EEG waves during anesthesia or undesirable deep periods in Bispectral index (BIS) monitoring on recovery agitation are the subject of this research.

DETAILED DESCRIPTION:
Many strategies have been developed to monitor perioperative anesthesia depth. Bispectral index (BIS) is a monitor that analyzes electroencephalogram (EEG) data and produces a numerical value. This value indicates the patient's level of consciousness and helps evaluate the depth of anesthesia. BIS is a routinely used monitor that continuously monitors the patient's state of consciousness during anesthesia. In this way, the depth of anesthesia can be controlled more precisely (1). When the level of consciousness is deep, the BIS value decreases and increases as the surface is approached. With this feature, it ensures that the patient's depth of anesthesia is kept at an optimal level and adjusted when necessary. This may help minimize anesthesia-related complications(2). BIS alone may not be sufficient to evaluate the depth of anesthesia. It should be used in conjunction with other clinical findings and monitors. Nowadays, anesthesia depth monitoring is a widely used method and is performed routinely in our clinic.

Many strategies have been developed to monitor perioperative anesthesia depth. BIS is a monitor that analyzes electroencephalogram (EEG) data and produces a numerical value. This value indicates the patient's level of consciousness and helps evaluate the depth of anesthesia. BIS is a routinely used monitor that continuously monitors the patient's state of consciousness during anesthesia. In this way, the depth of anesthesia can be controlled more precisely (1). When the level of consciousness is deep, the BIS value decreases and increases as the surface is approached. With this feature, it ensures that the patient's depth of anesthesia is kept at an optimal level and adjusted when necessary. This may help minimize anesthesia-related complications(2). BIS alone may not be sufficient to evaluate the depth of anesthesia. It should be used in conjunction with other clinical findings and monitors. Nowadays, anesthesia depth monitoring is a widely used method and is performed routinely in our clinic.

BIS (Bisspectral Index) Suppression Ratio is a value that measures the suppression rate of brain activity during anesthesia (3). This rate is calculated by analyzing EEG (Electroencephalogram) signals. This ratio indicates significant decreases in brain activity and increases as anesthesia deepens (4). Suppression is often desired in cases of deep anesthesia, especially during surgical intervention. However, an excessively high suppression rate can lead to delayed recovery times. The use of BIS Suppression Ratio in anesthesia management can help to more precisely control the patient's arousal process and the depth of general anesthesia. This value provides the anesthesia team with a guide to optimize the patient's state of consciousness and minimize complications that may occur during anesthesia. However, it is important that BIS Suppression Ratio should not be evaluated alone and should be used in conjunction with other clinical information(5). Each patient's response may be different, and therefore the anesthesia team must manage the depth of anesthesia by considering multiple factors. It has been shown in the literature that BIS Suppression Ratio (SR) values >40 have a similar effect to low BIS values. However, the undesirable Suppression Ratio in terms of number and duration is not fully known (6).

"Recovery agitation" generally refers to a situation that may occur after a surgical intervention or anesthesia. This condition describes the restlessness and agitation (symptoms such as restlessness, tension, insomnia) that the patient shows during the awakening process and during the recovery period from anesthesia. Recovery agitation sometimes occurs when the patient tries to wake up. It may occur when it starts and is usually a short-term condition that resolves on its own. However, in some cases, this agitation may be more pronounced and disturbing. This may affect the patient's condition and relaxation. The severity of the agitation may vary from person to person. Rapid recovery from anesthesia in the clinic is also a risk of agitation. Riker Sedation-Agitation Scale and Richmond Agitation-Sedation scale are the most frequently used methods to measure recovery agitation (7).

When the literature is examined, there are not enough studies on Bis suppression ratio and its relationship with recovery agitation is not yet known enough. For this purpose, our study aimed to question this relationship.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who will undergo lumbar disc herniation surgery in Kocaeli city hospital operating rooms will be included in our study after ethics committee approval.

  2. Patients over the age of 18 will be included in the study.

  3. Patients with an ASA score of 1-2 and without neurological disease will be included.

  4.Patients without known vascular diseases will be included.

  5. Study patients will receive routine anesthesia premedication and routine analgesics, and patients with different procedures will not be included in the study.

Exclusion Criteria:

* 1. Patients who do not want to participate in the study will not be included.

  2. Patients with intraoperative profound hypotension (mean arterial pressure <50) will be excluded.

  3. Those who develop intraoperative hypothermia or other anesthesia complications will be removed.

  4. Patients who will not be extubated postoperatively will be excluded from the study.

  5. Those with neurological diseases or using psychiatric medications will also be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The current research was designed as a prospective observational study. Routine anesthesia procedures will be applied to patients who will undergo lumbar disc herniation surgery and who have agreed to participate in the study, and the routinely recorded recovery scale will be recorded for the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
The relationship between BIS-SR values and post-anesthesia recovery (Richmond agitation sedation score) and recovery time | intraoperative period and postoperative first 4 hours
  The relationship between the maximum BIS-SR value or the time of SR>10 points and recovery times and recovery agitation (Richmond agitation sedation score) will be investigated.

SECONDARY OUTCOMES:
The relationship between Bis values and recovery agitation (Richmond agitation sedation score) | intraoperative period and postoperative first 4 hours
  A relationship between Bis values and recovery agitation (Richmond agitation sedation score) will be investigated. Possible changes in SR values will also be observed when BIS is in the range of 40-60 percent.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YUKSEK, Md, Study Chair — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
In case of appropriate request, anonymous patient results and raw data can be shared with written request and institutional permission.

REFERENCES:
- [Background] Cornelius BW, Jacobs TM. Pseudocholinesterase Deficiency Considerations: A Case Study. Anesth Prog. 2020 Sep 1;67(3):177-184. doi: 10.2344/anpr-67-03-16. PMID 32992329
- [Background] Eertmans W, Genbrugge C, Vander Laenen M, Boer W, Mesotten D, Dens J, Jans F, De Deyne C. The prognostic value of bispectral index and suppression ratio monitoring after out-of-hospital cardiac arrest: a prospective observational study. Ann Intensive Care. 2018 Mar 2;8(1):34. doi: 10.1186/s13613-018-0380-z. PMID 29500559
- [Background] Evered LA, Chan MTV, Han R, Chu MHM, Cheng BP, Scott DA, Pryor KO, Sessler DI, Veselis R, Frampton C, Sumner M, Ayeni A, Myles PS, Campbell D, Leslie K, Short TG. Anaesthetic depth and delirium after major surgery: a randomised clinical trial. Br J Anaesth. 2021 Nov;127(5):704-712. doi: 10.1016/j.bja.2021.07.021. Epub 2021 Aug 28. PMID 34465469
- [Background] Riker RR, Fraser GL, Wilkins ML. Comparing the bispectral index and suppression ratio with burst suppression of the electroencephalogram during pentobarbital infusions in adult intensive care patients. Pharmacotherapy. 2003 Sep;23(9):1087-93. doi: 10.1592/phco.23.10.1087.32766. PMID 14524640
- [Result] Kreuer S, Wilhelm W, Grundmann U, Larsen R, Bruhn J. Narcotrend index versus bispectral index as electroencephalogram measures of anesthetic drug effect during propofol anesthesia. Anesth Analg. 2004 Mar;98(3):692-7, table of contents. doi: 10.1213/01.ane.0000103182.78466.ef. PMID 14980921
- [Result] Selig C, Riegger C, Dirks B, Pawlik M, Seyfried T, Klingler W. Bispectral index (BIS) and suppression ratio (SR) as an early predictor of unfavourable neurological outcome after cardiac arrest. Resuscitation. 2014 Feb;85(2):221-6. doi: 10.1016/j.resuscitation.2013.11.008. Epub 2013 Nov 25. PMID 24287327